CLINICAL TRIAL: NCT03191734
Title: French Aquablation Clinical Investigation Using Waterjet Ablation Therapy for Endoscopic Resection of Prostate Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PROCEPT BioRobotics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP0112
Record Dates: First submitted 2017-06-13; First posted 2017-06-19 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
Keywords: Lower Urinary Tract Symptoms (LUTS); Benign Prostatic Hyperplasia (BPH); AQUABEAM; Aquablation
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AQUABEAM System (Experimental): AQUABEAM System
  Interventions: Device: AQUABEAM System

INTERVENTIONS:
Device: AQUABEAM System — Aquablation is a minimally invasive transurethral surgical procedure using the AQUABEAM system, a personalized image-guided waterject resection system that utilizes a high-pressure saline stream to resect and remove prostate tissue.

SUMMARY:
Single arm, multi-center prospective clinical trial to determine the safety and effectiveness of the AQUABEAM System in the treatment of benign prostatic hyperplasia (BPH) in men 45 to 80 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Subject has diagnosis of lower urinary tract symptoms due to benign prostatic enlargement causing bladder outlet obstruction.
* History of inadequate response, contraindication or refusal to medical therapy for BPH.
* Age from 45 through 80 years.
* Prostate volume between 30mL and 80mL by transrectal ultrasound (TRUS) measured at baseline.

Exclusion Criteria:

* BMI ≥ 42.
* IPSS total score <12.
* History of prostate cancer or clinically significant elevated PSA value.
* History of bladder cancer actively treated within 2 years prior to the surgical procedure.
* Bladder calculus or clinically significant bladder diverticulum (e.g., pouch size >20% of full bladder size).
* Active infection, including urinary tract infection within 72 hours of the treatment procedure.
* Prostatitis treated with antibiotics within 1 year of the surgical procedure.
* Subject ever diagnosed with urethral stricture, meatal stenosis, or bladder neck contracture, or has history of damage to external urinary sphincter.
* Subject has current diagnosis of stress urinary incontinence that requires treatment or daily pad or device use.
* Clinically significant abnormal serum creatinine measured within 30 days of treatment.
* Maximum urinary flow rate (Qmax) >15 mL/s or PVR > 300 mL measured by uroflowmetry test at baseline.
* Subject has been catheterized due to retention within 14 days prior to the surgical procedure.
* Subject has a history of intermittent self-catheterization.
* Previous prostate surgery or history of other lower urinary tract surgery such as e.g. urinary diversion, artificial urinary sphincter or penile prosthesis
* Subjects on anticoagulants or antiplatelet (if medication cannot be stopped before and after procedure) or known coagulopathy (except aspirin below 100mg/d)
* Any severe illness or psychiatric condition that would prevent study completion or confound study results.
* Subject taking systemic immune-suppressants including corticosteroids; unable to withhold non- steroidal anti-inflammatory agents (NSAIDs, including aspirin) for 3-5 days prior to treatment except for low dose aspirin (e.g. less than 100mg).
* Participants using medications specifically for bladder muscle problems (e.g., irritability). Use of medications with anticholinergic or similar properties is allowable provided the patient does not have documented adverse urinary side effects from these medications.
* Participating in another investigational study that could affect responses to the study device.
* Subject is unwilling to accept a transfusion should one be required.

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2019-01-07 (Actual)

PRIMARY OUTCOMES:
AQUABEAM System Effectiveness: IPSS total score change | 6 Months Post-op
  IPSS total score change from baseline to 6 Month

CONTACTS AND LOCATIONS:
Overall Officials: Aurelien Descazeaud, MD, Principal Investigator — Centre Hospitalier Régional Universitaire de Limoges
Locations (3):
- France (3):
  - CHU de Limoges, Limoges
  - Hôpital Cochin, Paris
  - Clinique Pasteur, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided